CLINICAL TRIAL: NCT04554511
Title: Prognostic Nomogram of Extranodal NK/T-cell Lymphoma: A Multi-center Retrospective Study
Brief Title: Prognostic Nomogram of Extranodal NK/T-cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, associate chief physician, Sun Yat-sen University
Other Study IDs: ENKTL-2020
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Patients diagnosed with ENKTL, between January 1, 2000 and August 31, 2020.
- Validation Cohort: Patients diagnosed with ENKTL, between January 1, 2000 and August 31, 2020.

SUMMARY:
This study aims to evaluate prognostic factors for overall survival and explore risk progression-free survival in ENKTL, and establish a prognostic predictive nomogram for ENKTL patients.

DETAILED DESCRIPTION:
This is a retrospective cohort study using anonymized information from patients with ENKTL. The following criteria are required: (1) Patients diagnosed with ENKTL between January 1, 2000 and August 31, 2020; (2) Patients older than 18 years. The pathology of initial diagnosis was reviewed by designated pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with ENKTL
* Patients diagnosed between January 1, 2000 and August 31, 2020
* Patients older than 18 years

Exclusion Criteria:

* Patients who did not have complete clinical information or immunohistochemistry, or who were lost follow-up immediately after treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients diagnosed with ENKTL, between January 1, 2000 and August 31, 2020;
  2. Patients older than 18 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year
  Time between the date of diagnosis and any kinds of death

SECONDARY OUTCOMES:
Progression-free survival | 5 year
  Time between the date of diagnosis and any kinds of death or relapse/progression

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China